CLINICAL TRIAL: NCT00720798
Title: Long-term Extension Study of Safety During Treatment With Tocilizumab (MRA) in Patients Completing Treatment in MRA Core Studies
Brief Title: An Extension Study of Tocilizumab (Myeloma Receptor Antibody [MRA]) in Patients Completing Treatment in Tocilizumab Core Studies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WA18696
Record Dates: First submitted 2008-07-22; First posted 2008-07-23 (Estimated); Results first posted 2014-09-30 (Estimated); Last update posted 2014-09-30 (Estimated); Status verified 2014-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab; Antirheumatic Agents; Adrenal Cortex Hormones

ARMS (1):
- Tocilizumab (Experimental): Participants received tocilizumab 8 mg/kg intravenously every 4 weeks till the end of the study (up to 7 years, 7 months). In addition, participants may have also received disease-modifying anti-rheumatic drugs, non-steroidal anti-inflammatory drugs, and oral corticosteroids at the discretion of the investigator.
  Interventions: Drug: Tocilizumab; Drug: Disease-modifying anti-rheumatic drugs; Drug: Non-steroidal anti-inflammatory drugs; Drug: Oral corticosteroids

INTERVENTIONS:
Drug: Tocilizumab — For participants weighing > 100 kg, the maximum dose of tocilizumab was 800 mg. Tocilizumab was supplied as a sterile solution in vials.
  Other Names: RoActemra; Actemra
Drug: Disease-modifying anti-rheumatic drugs — Disease-modifying anti-rheumatic drugs included methotrexate, chloroquine, hydroxychloroquine, parenteral gold, sulfasalazine, azathioprine, and leflunomide. These drugs could be used alone or in combination, except for the combination of methotrexate and leflunomide, which was not allowed.
Drug: Non-steroidal anti-inflammatory drugs — Participants could be treated with non-steroidal anti-inflammatory drugs up to the maximum recommended dose throughout the study. The choice and doses of non-steroidal anti-inflammatory drugs were at the discretion of the investigator.
Drug: Oral corticosteroids — Oral corticosteroids (≤ 10 mg/day) were permitted during the study.

SUMMARY:
This single-arm study evaluated the long-term efficacy and safety of tocilizumab in participants who had completed treatment in the tocilizumab core studies (NCT00106522 [Roche protocol WA18062], NCT00106574 [Roche protocol WA18063], and NCT00109408 [Roche protocol WA17824]) of adults with rheumatoid arthritis. Participants received tocilizumab alone or in combination with standard anti-rheumatic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have completed participation in 1 of the core studies in adult rheumatoid arthritis.

Exclusion Criteria:

* Treatment with any investigational agent since the last administration of study drug in the core studies.
* Treatment with iv gamma globulin, plasmapheresis, or prosorba column since the last administration of study drug in the core studies.
* Treatment with an anti-TNF or anti-IL1 agent, a T-cell co-stimulation modulator, or any biologic since the last administration of study drug in the core studies.
* Immunization with a live/attenuated vaccine since the last administration of study drug in the core studies.
* Previous treatment with any cell-depleting therapies, including investigational agents.
* Parenteral, intramuscular, or intra-articular corticosteroids within 6 weeks prior to baseline in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2067 (Actual)
Dates: Start 2005-09; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (261):
- United States (122):
  - Birmingham, Alabama
  - Huntsville, Alabama
  - Mesa, Arizona
  - Paradise Valley, Arizona
  - Peoria, Arizona
  - Scottsdale, Arizona
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Anaheim, California
  - Long Beach, California
  - Los Angeles, California
  - Palm Desert, California
  - Palm Springs, California
  - Palo Alto, California
  - San Diego, California
  - San Jose, California
  - San Leandro, California
  - Santa Maria, California
  - Torrance, California
  - Upland, California
  - Colorado Springs, Colorado
  - Newark, Delaware
  - Aventura, Florida
  - Delray Beach, Florida
  - Fort Lauderdale, Florida
  - Palm Habor, Florida
  - Palm Harbor, Florida
  - Sarasota, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Boise, Idaho
  - Idaho Falls, Idaho
  - Meridian, Idaho
  - Morton Grove, Illinois
  - Springfield, Illinois
  - Vernon Hills, Illinois
  - Indianapolis, Indiana
  - Cedar Rapids, Iowa
  - Des Moines, Iowa
  - Bowling Green, Kentucky
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Baton Rouge, Louisiana
  - Shreverport, Louisiana
  - Slidell, Louisiana
  - Portland, Maine
  - Frederick, Maryland
  - Wheaton, Maryland
  - Boston, Massachusetts
  - Pittsfield, Massachusetts
  - Grand Rapids, Michigan
  - Kalamazoo, Michigan
  - Lansing, Michigan
  - Eagan, Minnesota
  - Saint Cloud, Minnesota
  - Saint Louis Park, Minnesota
  - Flowood, Mississippi
  - Tupelo, Mississippi
  - Springfield, Missouri
  - St Louis, Missouri
  - Billings, Montana
  - Lincoln, Nebraska
  - Reno, Nevada
  - Dover, New Hampshire
  - Haddon Heights, New Jersey
  - New Brunswick, New Jersey
  - Passaic, New Jersey
  - Albuquerque, New Mexico
  - Albany, New York
  - Binghamton, New York
  - Great Neck, New York
  - New York, New York
  - Orchard Park, New York
  - Plainview, New York
  - Rochester, New York
  - Syracuse, New York
  - Asheville, North Carolina
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Raleigh, North Carolina
  - Bismarck, North Dakota
  - Canton, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Dayton, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Eugene, Oregon
  - Medford, Oregon
  - Allentown, Pennsylvania
  - Bethlehem, Pennsylvania
  - Danville, Pennsylvania
  - Duncansville, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Willow Grove, Pennsylvania
  - Wyomissing, Pennsylvania
  - Johnston, Rhode Island
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Greenville, South Carolina
  - Hickory Grove, South Carolina
  - Hixson, Tennessee
  - Jackson, Tennessee
  - Nashville, Tennessee
  - Amarillo, Texas
  - Austin, Texas
  - Dallas, Texas
  - Houston, Texas
  - Mesquite, Texas
  - Burlington, Vermont
  - Chesapeake, Virginia
  - Norfolk, Virginia
  - Mountlake Terrace, Washington
  - Olympia, Washington
  - Seattle, Washington
  - Spokane, Washington
  - Tacoma, Washington
  - Glendale, Wisconsin
  - La Crosse, Wisconsin
- Argentina (3):
  - Buenos Aires
  - Rosario
  - San Juan Bautista
- Australia (5):
  - Hobart
  - Malvern
  - Shenton Park
  - Sydney
  - Woolloongabba
- Belgium (2):
  - Hasselt
  - Merksem
- Brazil (3):
  - Campinas
  - Goiânia
  - Rio de Janeiro
- Canada (16):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Victoria, British Columbia
  - Winnipeg, Manitoba
  - St. John's, Newfoundland and Labrador
  - Burlington, Ontario
  - Hamilton, Ontario
  - Kitchener, Ontario
  - London, Ontario
  - Mississauga, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Québec, Quebec
  - Sainte-Foy, Quebec
  - Saskatoon, Saskatchewan
- China (5):
  - Beijing
  - Guangzhou
  - Hefei Anhui
  - Jinan
  - Shanghai
- San José, Costa Rica
- Czechia (2):
  - Hradec Králové
  - Prague
- Hellerup, Denmark
- Finland (2):
  - Helsinki
  - Jyväskylä
- France (19):
  - Amiens
  - Bordeaux
  - Boulogne-Billancourt
  - Brest
  - Grenoble
  - Le Kremlin-Bicêtre
  - Lille
  - Lyon
  - Marseille
  - Montpellier
  - Nantes
  - Nice
  - Paris
  - Pierre-Bénite
  - Rennes
  - Rouen
  - Saint-Priest-en-Jarez
  - Strasbourg
  - Toulouse
- Germany (13):
  - Aachen
  - Berlin
  - Cologne
  - Dresden
  - Essen
  - Gommern
  - Herne
  - Hildesheim
  - München
  - Osnabrück
  - Sendenhorst
  - Wiesbaden
  - Würzburg
- Hong Kong (2):
  - Hong Kong
  - Tuenmen
- Reykjavik, Iceland
- Israel (3):
  - Ashkelon
  - Haifa
  - Rishon LeZiyyon
- Italy (8):
  - Brescia
  - Genova
  - Milan
  - Padua
  - Pavia
  - Pisa
  - Siena
  - Udine
- Lithuania (5):
  - Kaunas
  - Klaipėda
  - Panevezys
  - Šiauliai
  - Vilnius
- Mexico (4):
  - Guadalajara
  - León
  - Mexico City
  - Tijuana
- Nijmegen, Netherlands
- Norway (2):
  - Levanger
  - Lillehammer
- Panama City, Panama
- Lima, Peru
- Lisbon, Portugal
- Ponce, Puerto Rico
- Russia (4):
  - Moscow
  - Ryazan
  - Saint Petersburg
  - Tula
- Serbia (2):
  - Belgrade
  - Niška Banja
- Slovenia (2):
  - Ljubljana
  - Maribor
- South Africa (6):
  - Cape Town
  - Diepkloof
  - Durban
  - Pinelands
  - Pretoria
  - Radiokop
- Spain (6):
  - Barakaldo
  - Barcelona
  - Madrid
  - Málaga
  - Pontevedra
  - Santiago de Compostela
- Sweden (2):
  - Stockholm
  - Umeå
- Lausanne, Switzerland
- Thailand (2):
  - Bangkok
  - Chiang Mai
- United Kingdom (12):
  - Basingstoke
  - Birmingham
  - Cannock
  - Derby
  - Leeds
  - London
  - Manchester
  - Middlesbrough
  - Newcastle upon Tyne
  - Oxford
  - Southampton
  - Stoke-on-Trent

REFERENCES:
- [Derived] Jones G, Wallace T, McIntosh MJ, Brockwell L, Gomez-Reino JJ, Sebba A. Five-year Efficacy and Safety of Tocilizumab Monotherapy in Patients with Rheumatoid Arthritis Who Were Methotrexate- and Biologic-naive or Free of Methotrexate for 6 Months: the AMBITION Study. J Rheumatol. 2017 Feb;44(2):142-146. doi: 10.3899/jrheum.160287. Epub 2016 Dec 1. PMID 27909081

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tocilizumab
Started | 2067
Completed | 1311
Not Completed | 756
Not completed — Adverse Event | 304
Not completed — Death | 39
Not completed — Insufficient Therapeutic Response | 129
Not completed — Protocol Violation | 4
Not completed — Refused Treatment | 151
Not completed — Failure to Return | 46
Not completed — Reason not Specified | 83

BASELINE CHARACTERISTICS:
Population: All-exposure population: All participants who entered this study and received at least 1 dose of tocilizumab in either this extension study or in a core study.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 2067
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.2 (12.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1689
  Male | 378

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With ≥ 1 Adverse Event
Time Frame: Baseline to the end of the study (up to 7 years, 7 months)
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 2067
Percentage of participants | 96.3

2. Secondary Outcome: Percentage of Participants Who Withdrew From Treatment
Time Frame: Baseline to the end of the study (up to 7 years, 7 months)
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 2067
Percentage of participants | 36.6

3. Secondary Outcome: Percentage of Participants With Concomitant Oral Corticosteroid Therapy
Description: Concomitant therapy with oral corticosteroids (up 5 to 10 mg daily prednisone or equivalent) was permitted in the study. Reduction of oral corticosteroids was permitted, but not required, if a patient achieved at least a 50% improvement from baseline in both tender joint count and swollen joint count.
  The data are reported for each 6-month period of the study where a month = 28 days. The last 6-month period is for months 96 through 101. The actually study duration in 28-day months was 98.85 months.
Time Frame: Baseline to the end of the study (up to 7 years, 7 months)
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 2067
Percentage of participants
  0 - 6 Months, n = 2067 | 55.8
  6 - 12 Months, n = 2041 | 55.3
  12 - 18 Months, n = 1944 | 54.6
  18 - 24 Months, n = 1832 | 54.3
  24 - 30 Months, n = 1753 | 53.2
  30 - 36 Months, n = 1677 | 52.9
  36 - 42 Months, n = 1620 | 51.3
  42 - 48 Months, n = 1568 | 50.4
  48 - 54 Months, n = 1516 | 50.6
  54 - 60 Months, n = 1475 | 50.1
  60 - 66 Months, n = 1423 | 49.2
  66 - 72 Months, n = 1342 | 48.4
  72 - 78 Months, n = 788 | 48.7
  78 - 84 Months, n = 62 | 72.6
  84 - 90 Months, n = 34 | 79.4
  90 - 96 Months, n = 10 | 70.0
  96 - 102 Months, n = 2 | 0.0

4. Secondary Outcome: Percentage of Participants Who Changed From Monotherapy to Combination Therapy
Description: Participants who entered this study from study WA17824 on tocilizumab monotherapy, who did not achieve a 50% reduction in tender and swollen joint counts from Baseline of study WA17824, could add methotrexate or another allowable disease-modifying anti-rheumatic drug, according to the investigator's practice and as tolerated by the patient, at any time during this study.
Time Frame: Baseline to Week 296
Population: All-exposure population: All participants who entered this study and received at least 1 dose of tocilizumab in either this extension study or in a core study. Only participants from the core study WA17824 are included in the analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 243
Percentage of participants
  Week 8 | 1.2
  Week 12 | 0.4
  Week 24 | 15.6
  Week 28 | 7.0
  Week 32 | 2.5
  Week 36 | 1.6
  Week 40 | 0.4
  Week 44 | 0.4
  Week 48 | 1.6
  Week 52 | 0.8
  Week 54 | 0.8
  Week 64 | 1.2
  Week 68 | 0.8
  Week 72 | 0.8
  Week 76 | 0.4
  Week 88 | 0.8
  Week 96 | 1.2
  Week 100 | 0.8
  Week 104 | 0.4
  Week 108 | 0.4
  Week 112 | 0.4
  Week 116 | 0.4
  Week 120 | 0.4
  Week 140 | 0.4
  Week 152 | 0.8
  Week 184 | 0.4
  Week 196 | 0.4
  Week 200 | 0.8
  Week 292 | 0.4
  Week 296 | 0.8

5. Secondary Outcome: Percentage of Participants With an Improvement of at Least 20%, 50%, 70%, or 90% in the American College of Rheumatology (ACR) Score (ACR20/50/70/90) From Baseline at Weeks 24, 48, 108, 156, 204, and 264
Description: Improvement must be seen in tender (68 assessed joints) and swollen joint counts (66 assessed joints) and in at least 3 of the following 5 parameters: Separate patient and physician assessments of patient disease activity in the previous 24 hours on a visual analog scale (VAS, the left end of the scale "no disease activity" [symptom-free and no arthritis symptoms], right end of the scale "maximum disease activity"); patient assessment of pain in the previous 24 hours on a VAS (left end of the scale "no pain", right end of the scale "unbearable pain"); Health Assessment Questionnaire-Disability Index (20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities, 0=without difficulty to 3=unable to do); and erythrocyte sedimentation rate.
Time Frame: Baseline to Week 264
Population: All-exposure population: All participants who entered this study and received at least 1 dose of tocilizumab in either this extension study or in a core study. Only participants with available data were included in the analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 2067
Percentage of participants
  ACR20 Week 24 (n=1966) | 59.5
  ACR20 Week 48 (n=1825) | 66.7
  ACR20 Week 108 (n=1607) | 74.1
  ACR20 Week 156 (n=1512) | 74.3
  ACR20 Week 204 (n=1415) | 77.5
  ACR20 Week 264 (n = 1319) | 78.7
  ACR50 Week 24 (n=1966) | 34.9
  ACR50 Week 48 (n=1825) | 44.4
  ACR50 Week 108 (n=1607) | 52.8
  ACR50 Week 156 (n=1512) | 54.7
  ACR50 Week 204 (n=1415) | 56.5
  ACR50 Week 264 (n= 1319) | 58.8
  ACR70 Week 24 (n=1966) | 17.8
  ACR70 Week 48 (n=1825) | 25.5
  ACR70 Week 108 (n=1607) | 33.2
  ACR70 Week 156 (n=1512) | 35.7
  ACR70 Week 204 (n =1415) | 38.6
  ACR70 Week 264 (n=1319) | 40.5
  ACR90 Week 24 (n=1966) | 4.3
  ACR90 Week 48 (n=1825 | 7.9
  ACR90 Week 108 (n=1607) | 12.1
  ACR90 Week 156 (n=1512) | 14.7
  ACR90 Week 204 (n=1415) | 17.7
  ACR90 Week 264 (n=1319) | 18.1

6. Secondary Outcome: Percentage of Participants Who Achieved a Major Clinical Response at Weeks 48, 96, 144, 192, and 264
Description: A major clinical response was defined as maintenance of an improvement of at least 70% in the American College of Rheumatology (ACR) score (ACR70) for at least 24 weeks. Improvement must be seen in tender (68 assessed joints) and swollen joint counts (66 assessed joints) and in at least 3 of the following 5 parameters: Separate patient and physician assessments of patient disease activity in the previous 24 hours on a visual analog scale (VAS, the left end of the scale "no disease activity" [symptom-free and no arthritis symptoms], right end of the scale "maximum disease activity"); patient assessment of pain in the previous 24 hours on a VAS (left end of the scale "no pain", right end of the scale "unbearable pain"); Health Assessment Questionnaire-Disability Index (20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities, 0=without difficulty to 3=unable to do); and erythrocyte sedimentation rate.
Time Frame: Baseline to Week 264
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 2067
Percentage of participants
  Week 48 (n = 1937) | 8.5
  Week 96 (n = 1745) | 16.2
  Week 144 (n = 1615) | 20.9
  Week 192 (n = 1514) | 22.9
  Week 264 (n = 1358) | 24.9

7. Secondary Outcome: Percentage of Participants Who Maintained an Improvement of at Least 20%, 50%, or 70% in the American College of Rheumatology (ACR) Score (ACR20/50/70) Consecutively for 24, 48, 96, and 264 Weeks at Weeks 48, 96, 144, 192, and 264
Description: as for outcome 5
Time Frame: Baseline to Week 264
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 2067
Percentage of participants
  ACR20 Week 48: Maintained 24 weeks (n=1937) | 41.2
  ACR20 Week 96: Maintained 24 weeks (n=1745) | 53.0
  ACR20 Week 96: Maintained 48 weeks (n=1745) | 43.0
  ACR20 Week 144: Maintained 24 weeks (n=1615) | 56.3
  ACR20 Week 144: Maintained 48 weeks (n=1615) | 48.7
  ACR20 Week 144: Maintained 96 weeks (n=1615) | 35.6
  ACR20 Week 192: Maintained 24 weeks (n=1514) | 60.0
  ACR20 Week 192: Maintained 48 weeks (n=1514) | 52.3
  ACR20 Week 192: Maintained 96 weeks (n=1514) | 41.3
  ACR20 Week 192: Maintained 144 weeks (n=1514) | 31.8
  ACR20 Week 264: Maintained 24 weeks (n=1358) | 63.0
  ACR20 Week 264: Maintained 48 weeks (n=1358) | 54.7
  ACR20 Week 264: Maintained 96 weeks (n=1358) | 46.2
  ACR20 Week 264: Maintained 144 weeks (n=1358) | 38.7
  ACR20 Week 264: Maintained 192 weeks (n=1358) | 32.6
  ACR50 Week 48: Maintained 24 weeks (n=1937) | 20.7
  ACR50 Week 96: Maintained 24 weeks (n=1745) | 32.0
  ACR50 Week 96: Maintained 48 weeks (n=1745) | 22.8
  ACR50 Week 144: Maintained 24 weeks (n=1615) | 36.9
  ACR50 Week 144: Maintained 48 weeks (n=1615) | 28.4
  ACR50 Week 144: Maintained 96 weeks (n=1615) | 18.1
  ACR50 Week 192: Maintained 24 weeks (n=1514) | 39.8
  ACR50 Week 192: Maintained 48 weeks (n=1514) | 33.0
  ACR50 Week 192: Maintained 96 weeks (n=1514) | 22.7
  ACR50 Week 192: Maintained 144 weeks (n=1514) | 15.9
  ACR50 Week 264: Maintained 24 weeks (n=1358) | 42.3
  ACR50 Week 264: Maintained 48 weeks (n=1358) | 34.7
  ACR50 Week 264: Maintained 96 weeks (n=1358) | 27.6
  ACR50 Week 264: Maintained 144 weeks (n=1358) | 21.7
  ACR50 Week 264: Maintained 192 weeks (n=1358) | 16.6
  ACR70 Week 48: Maintained 24 weeks (n=1937) | 8.5
  ACR70 Week 96: Maintained 24 weeks (n=1745) | 16.2
  ACR70 Week 96: Maintained 48 weeks (n=1745) | 11.2
  ACR70 Week 144: Maintained 4 weeks (n=1615) | 20.9
  ACR70 Week 144: Maintained 48 weeks (n=1615) | 15.0
  ACR70 Week 144: Maintained 96 weeks (n=1615) | 8.7
  ACR70 Week 192: Maintained 24 weeks (n=1514) | 22.9
  ACR70 Week 192: Maintained 48 weeks (n=1514) | 17.6
  ACR70 Week 192: Maintained 96 weeks (n=1514) | 11.4
  ACR70 Week 192: Maintained 144 weeks (n=1514) | 7.3
  ACR70 Week 264: Maintained 24 weeks (n=1358) | 24.9
  ACR70 Week 264: Maintained 48 weeks (n=1358) | 19.7
  ACR70 Week 264: Maintained 96 weeks (n=1358) | 14.4
  ACR70 Week 264: Maintained 144 weeks (n=1358) | 11.0
  ACR70 Week 264: Maintained 192 weeks (n=1358) | 7.7

8. Secondary Outcome: Swollen and Tender Joint Count (SJC/TJC) at Baseline and Weeks 24, 48, 108, 156, 204, and 264
Description: The number of swollen (66 assessed joints) and tender (68 assessed joints) joints was assessed. Joints were physically examined and classified as swollen/not swollen and tender/not tender by pressure and joint manipulation.
Time Frame: Baseline to Week 264
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | Tocilizumab
Number analyzed (Participants) | 2067
Joints
  Baseline SJC (n = 2047) | 17.4 (11.96)
  Week 24 SJC (n = 2010) | 8.2 (9.43)
  Week 48 SJC (n = 1924) | 6.4 (8.75)
  Week 108 SJC (n = 1692) | 4.2 (6.69)
  Week 156 SJC (n = 1580) | 4.0 (7.09)
  Week 204 SJC (n = 1482) | 3.2 (5.96)
  Week 264 SJC (n = 1352) | 2.9 (5.85)
  Baseline TJC (n = 2047) | 27.3 (16.97)
  Week 24 TJC (n = 2010) | 12.8 (14.10)
  Week 48 TJC (n = 1924) | 10.3 (12.99)
  Week 108 TJC (n = 1692) | 7.8 (11.04)
  Week 156 TJC (n = 1580) | 7.2 (11.03)
  Week 204 TJC (n = 1482) | 6.1 (9.83)
  Week 264 TJC (n = 1352) | 5.6 (9.48)

9. Secondary Outcome: Disease Activity and Pain at Baseline and Weeks 24, 48, 108, 156, 204, and 264
Description: Participant's made a global assessment of their current disease activity on a 100 mm horizontal visual analogue scale (VAS). The left end of the scale indicated "no disease activity" (symptom-free and no arthritis symptoms, score = 0) and the right end indicated "maximum disease activity" (maximum arthritis disease activity, score = 100). The participant's treating physician made a global assessment of the participant's current disease activity on a 100 mm horizontal VAS. The left end of the scale indicated "no disease activity" (symptom-free and no arthritis symptoms, score = 0) and the right end indicated "maximum disease activity" (maximum arthritis disease activity, score = 100). Participant's made an assessment of their current level of pain on a 100 mm horizontal VAS. The left end of the scale indicated "no pain" (score = 0) and the right end of the scale indicated "unbearable pain" (score = 100).
Time Frame: Baseline to Week 264
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab
Number analyzed (Participants) | 2067
mm
  Participant Disease Activity - Baseline (n=2039) | 60.5 (25.52)
  Participant Disease Activity - Week 24 (n=1989) | 34.4 (26.03)
  Participant Disease Activity - Week 48 (n=1840) | 31.7 (25.25)
  Participant Disease Activity - Week 108 (n=1621) | 29.2 (24.75)
  Participant Disease Activity - Week 156 (n=1515) | 28.5 (25.16)
  Participant Disease Activity - Week 204 (n=1427) | 27.4 (24.72)
  Participant Disease Activity - Week 264 (n=1328) | 27.4 (25.50)
  Physician Disease Activity - Baseline (n=2043) | 57.3 (22.04)
  Physician Disease Activity - Week 24 (n=1990) | 26.8 (20.22)
  Physician Disease Activity - Week 48 (n=1830) | 22.3 (18.93)
  Physician Disease Activity - Week 108 (n=1619) | 18.6 (17.59)
  Physician Disease Activity - Week 156 (n=1516) | 17.4 (17.21)
  Physician Disease Activity - Week 204 (n=1413) | 15.6 (16.49)
  Physician Disease Activity - Week 264 (n=1330) | 15.1 (16.51)
  Participant Pain - Baseline (n=2041) | 54.9 (25.00)
  Participant Pain - Week 24 (n=1991) | 31.0 (24.56)
  Participant Pain - Week 48 (n=1842) | 28.0 (23.76)
  Participant Pain - Week 108 (n=1622) | 26.6 (23.52)
  Participant Pain - Week 156 (n=1517) | 26.2 (23.90)
  Participant Pain - Week 204 (n=1428) | 25.3 (23.05)
  Participant Pain - Week 264 (n=1329) | 25.1 (23.72)

10. Secondary Outcome: Health Assessment Questionnaire-Disability Index Score at Baseline and Weeks 24, 48, 108, 156, 204, and 264
Description: The Health Assessment Questionnaire-Disability Index (HAQ-DI), as a measure of functional ability, consists of 30 questions in 8 domains: Dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities. There are 4 possible responses to each question (0=without any difficulty, 1=with some difficulty, 2=with much difficulty, 3=unable to do). A domain score is the highest score in that domain. To calculate the overall score, the patient must have a domain score in at least 6 of the 8 domains. The HAQ-DI score is the sum of the domain scores divided by the number of domains that have a non-missing score and ranges from 0 (best) to 3 (worst). A higher score indicates less ability.
Time Frame: Baseline to Week 264
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 2067
Units on a scale
  Baseline (n = 2037) | 1.46 (0.660)
  Week 24 (n = 2008) | 1.04 (0.692)
  Week 48 (n = 1853) | 0.97 (0.693)
  Week 108 (n = 1635) | 0.89 (0.694)
  Week 156 (n = 1529) | 0.87 (0.689)
  Week 204 (n = 1438) | 0.84 (0.684)
  Week 264 (n = 1334) | 0.86 (0.696)

11. Secondary Outcome: Erythrocyte Sedimentation Rate at Baseline and Weeks 24, 48, 108, 156, 204, and 264
Description: Erythrocyte sedimentation rate (ESR) was determined locally.
Time Frame: Baseline to Week 264
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mm/h
Arm/Group | Tocilizumab
Number analyzed (Participants) | 2067
mm/h
  Baseline (n = 2047) | 46.2 (27.45)
  Week 24 (n = 1992) | 11.3 (14.97)
  Week 48 (n = 1830) | 10.2 (13.94)
  Week 108 (n = 1606) | 9.0 (12.79)
  Week 156 (n = 1509) | 8.9 (12.44)
  Week 204 (n = 1412) | 8.9 (12.01)
  Week 264 (n = 1329) | 9.7 (13.51)

12. Secondary Outcome: Change in the Disease Activity Score 28 (DAS-28) From Baseline to Weeks 24, 48, 96, and 264
Description: The DAS28 is a combined index for measuring disease activity in rheumatic arthritis (RA) and includes swollen and tender joint counts, erythrocyte sedimentation rate (ESR), and general health (GH) status. The index is calculated with the following formula: DAS28 = (0.56 × √(TJC28)) + (0.28 × √(SJC28)) + (0.7 × log(ESR)) + (0.014 × GH), where TJC28 = tender joint count and SJC28 = swollen joint count, each on 28 joints. GH = a patient's global assessment of disease activity in the previous 24 hours on a 100 mm visual analog scale (left end = no disease activity [symptom-free and no arthritis symptoms], right end = maximum disease activity [maximum arthritis disease activity]). When ESR equaled 0 mm/hr, it was set to 1 mm/hr. The DAS28 scale ranges from 0 to 10, where higher scores represent higher disease activity. A negative change score indicates improvement.
Time Frame: Baseline to Week 264
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 2067
Units on a scale
  Week 24 (n = 1920) | -2.82 (1.559)
  Week 48 (n = 1753) | -3.20 (1.644)
  Week 96 (n = 1596) | -3.46 (1.715)
  Week 264 (n = 1278) | -3.73 (1.742)

13. Secondary Outcome: Percentage of Participants Who Were Disease Activity Score 28 (DAS-28) Responders at Weeks 24, 48, 108, 156, 204, and 264
Description: A DAS-28 responder was defined as someone who met the European League Against Rheumatism [EULAR] criteria of a good or moderate response. A change of the DAS-28 score from Baseline was used to determine EULAR responses of good, moderate, or no response. For a post-baseline score ≤ 3.2, a change from baseline of < -1.2 was a good response, < -0.6 to ≥ -1.2 was a moderate response, and ≥ -0.6 was no response. For a post-baseline score > 3.2 to ≤ 5.1, a change from baseline of < -0.6 was a moderate response and ≥ -0.6 was no response. For a post-baseline score > 5.1, a change from baseline < -1.2 was a moderate response and ≥ -1.2 was no response. A good response could not be achieved for post-baseline scores > 3.2.
Time Frame: Baseline to Week 264
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 2067
Percentage of participants
  Week 24 Good (n = 1920) | 43.3
  Week 48 Good (n = 1753) | 51.9
  Week 108 Good (n = 1525) | 61.1
  Week 156 Good (n = 1441) | 64.7
  Week 204 Good (n = 1358) | 67.8
  Week 264 Good (n = 1278) | 68.8
  Week 24 Moderate (n = 1920) | 45.1
  Week 48 Moderate (n = 1753) | 40.0
  Week 108 Moderate (n = 1525) | 33.2
  Week 156 Moderate (n = 1441) | 28.7
  Week 204 Moderate (n = 1358) | 26.4
  Week 264 Moderate (n = 1278) | 26.1

14. Secondary Outcome: Percentage of Participants Who Maintained a Disease Activity Score 28 (DAS-28) Response for 24, 48, 96, 144, and 192 Weeks at Weeks 48, 96, 144, 192, and 264
Description: as for outcome 13
Time Frame: Baseline to Week 264
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 2067
Percentage of participants
  Week 48: Maintained response 24 weeks (n=1937) | 67.6
  Week 96: Maintained response 24 weeks (n=1745) | 72.7
  Week 96: Maintained response 48 weeks (n=1745) | 63.4
  Week 144: Maintained response 24 weeks (n=1615) | 73.1
  Week 144: Maintained response 48 weeks (n=1615) | 64.1
  Week 144: Maintained response 96 weeks (n=1615) | 52.9
  Week 192: Maintained response 24 weeks (n=1514) | 73.3
  Week 192: Maintained response 48 weeks (n=1514) | 64.7
  Week 192: Maintained response 96 weeks (n=1514) | 53.6
  Week 192: Maintained response 144 weeks (n=1514) | 45.5
  Week 264: Maintained response 24 weeks (n = 1358) | 76.7
  Week 264: Maintained response 48 weeks (n = 1358) | 68.6
  Week 264: Maintained response 96 weeks (n = 1358) | 56.4
  Week 264: Maintained response 144 weeks (n = 1358) | 48.7
  Week 264: Maintained response 192 weeks (n = 1358) | 42.1

15. Secondary Outcome: Percentage of Participants With a Clinically Relevant Improvement in Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) Score at Weeks 24, 36, 48, 108, 156, 204, and 264
Description: The FACIT-F is a 13-item participant self-report questionnaire that assesses fatigue over the previous 7 days by scoring each item on a 5-point scale (0=Not at all, 1=A little bit, 2=Somewhat, 3=Quite a bit, 4=Very much). An overall FACIT-F score was obtained by summing the scores of all 13 items. The overall score ranged from 0 to 52. A lower score indicates less fatigue. A clinically relevant improvement in the FACIT-F score was defined as a ≥ 5-point increase from Baseline.
Time Frame: Baseline to Week 264
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 2067
Percentage of participants
  Week 24 (n = 1984) | 59.5
  Week 36 (n = 1839) | 52.5
  Week 48 (n = 1803) | 56.0
  Week 108 (n = 1616) | 56.8
  Week 156 (n = 1513) | 56.3
  Week 204 (n = 1422) | 56.4
  Week 264 (n = 1320) | 61.9

16. Secondary Outcome: Percentage of Participants With a Clinically Relevant Improvement in the Physical and Mental Component Scores of the Short Form 36 (SF-36) Health Survey at Weeks 24, 48, 108, 156, 204, and 264
Description: The SF-36 Health Survey uses participant-reported symptoms on 8 subscales to assess health-related quality of life (HRQoL). The Physical Component Summary (PCS) score summarizes the subscales Physical Functioning, Role-Physical, Bodily Pain, and General Health. The Mental Component Summary (MCS) score summarizes the subscales Vitality, Social Functioning, Role-Emotional, and Mental Health. Each score was scaled from 0 to 100 with a higher score indicating better HRQoL. A clinically relevant improvement in the Physical and Mental Component Scores of the SF-36 was defined as a ≥ 5-point increase from Baseline.
Time Frame: Baseline to Week 264
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 2067
Percentage of participants
  Week 24 Mental Score (n = 1850) | 42.4
  Week 48 Mental Score (n = 1789) | 44.4
  Week 108 Mental Score (n = 1551) | 45.3
  Week 156 Mental Score (n = 1468) | 46.1
  Week 204 Mental Score (n = 1377) | 47.1
  Week 264 Mental Score (n = 1302) | 44.9
  Week 24 Physical Score (n = 1850) | 56.2
  Week 48 Physical Score (n = 1789) | 61.4
  Week 108 Physical Score (n = 1551) | 63.2
  Week 156 Physical Score (n = 1468) | 62.5
  Week 204 Physical Score (n = 1377) | 64.1
  Week 264 Physical Score (n = 1302) | 63.7

ADVERSE EVENTS:
Description: All-exposure population: All participants who entered this study and received at least 1 dose of tocilizumab in either this extension study or in a core study.
Arm/Group | Tocilizumab
Serious Adverse Events (participants affected / at risk) | 727/2067
Other Adverse Events (participants affected / at risk) | 1836/2067
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=2067)
Pneumonia (Infections and infestations) | 70
Cellulitis (Infections and infestations) | 57
Appendicitis (Infections and infestations) | 11
Diverticulitis (Infections and infestations) | 10
Gastroenteritis (Infections and infestations) | 10
Sepsis (Infections and infestations) | 10
Urinary tract infection (Infections and infestations) | 10
Arthritis bacterial (Infections and infestations) | 8
Bronchitis (Infections and infestations) | 7
Herpes zoster (Infections and infestations) | 7
Abscess limb (Infections and infestations) | 6
Erysipelas (Infections and infestations) | 6
Septic shock (Infections and infestations) | 6
Bronchopneumonia (Infections and infestations) | 5
Postoperative wound infection (Infections and infestations) | 5
Pyelonephritis (Infections and infestations) | 5
Infectious pleural effusion (Infections and infestations) | 4
Peritonitis (Infections and infestations) | 4
Pulmonary tuberculosis (Infections and infestations) | 4
Staphylococcal infection (Infections and infestations) | 4
Wound infection (Infections and infestations) | 4
Abdominal abscess (Infections and infestations) | 3
Bursitis infective (Infections and infestations) | 3
Staphylococcal Clostridium difficile colitis (Infections and infestations) | 3
Empyema (Infections and infestations) | 3
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 3
Lung infection (Infections and infestations) | 3
Necrotising fasciitis (Infections and infestations) | 3
Osteomyelitis (Infections and infestations) | 3
Pneumonia pneumococcal (Infections and infestations) | 3
Pneumonia staphylococcal (Infections and infestations) | 3
Post procedural infection (Infections and infestations) | 3
Septic arthritis (Infections and infestations) | 3
Staphylococcal sinusitis (Infections and infestations) | 3
Subcutaneous abscess (Infections and infestations) | 3
Wound infection staphylococcal (Infections and infestations) | 3
Abdominal wall abscess (Infections and infestations) | 2
Gastroenteritis viral (Infections and infestations) | 2
Infective tenosynovitis (Infections and infestations) | 2
Influenza (Infections and infestations) | 2
Liver abscess (Infections and infestations) | 2
Localised infection (Infections and infestations) | 2
Lower respiratory tract infection (Infections and infestations) | 2
Pelvic inflammatory disease (Infections and infestations) | 2
Pericolic abscess (Infections and infestations) | 2
Peritonitis bacterial (Infections and infestations) | 2
Pneumonia haemophilus (Infections and infestations) | 2
Pneumonia streptococcal (Infections and infestations) | 2
Pulmonary sepsis (Infections and infestations) | 2
Respiratory tract infection (Infections and infestations) | 2
Salmonellosis (Infections and infestations) | 2
Septic arthritis streptococcal (Infections and infestations) | 2
Sinusitis fungal (Infections and infestations) | 2
Soft tissue infection (Infections and infestations) | 2
Staphylococcal abscess (Infections and infestations) | 2
Tooth infection (Infections and infestations) | 2
Tuberculous pleurisy (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 2
Urosepsis (Infections and infestations) | 2
Viral infection (Infections and infestations) | 2
Abscess (Infections and infestations) | 1
Abscess oral (Infections and infestations) | 1
Abscess soft tissue (Infections and infestations) | 1
Acquired immunodeficiency syndrome (Infections and infestations) | 1
Alcaligenes infection (Infections and infestations) | 1
Anal abscess (Infections and infestations) | 1
Appendiceal abscess (Infections and infestations) | 1
Arthritis infective (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 1
Bacterial sepsis (Infections and infestations) | 1
Biliary sepsis (Infections and infestations) | 1
Breast abscess (Infections and infestations) | 1
Bronchitis bacterial (Infections and infestations) | 1
Bronchitis viral (Infections and infestations) | 1
Bursitis infective (Infections and infestations) | 1
Campylobacter gastroenteritis (Infections and infestations) | 1
Cellulitis gangrenous (Infections and infestations) | 1
Cellulitis staphylococcal (Infections and infestations) | 1
Central nervous system infection (Infections and infestations) | 1
Chronic tonsillitis (Infections and infestations) | 1
Encephalitis viral (Infections and infestations) | 1
Endocarditis bacterial (Infections and infestations) | 1
Endocarditis enterococcal (Infections and infestations) | 1
Enterocolitis infectious (Infections and infestations) | 1
Escherichia infection (Infections and infestations) | 1
Escherichia sepsis (Infections and infestations) | 1
Escherichia urinary tract infection (Infections and infestations) | 1
Extradural abscess (Infections and infestations) | 1
Fallopian tube abscess (Infections and infestations) | 1
Furuncle (Infections and infestations) | 1
Gingival infection (Infections and infestations) | 1
Haematoma infection (Infections and infestations) | 1
Hepatitis B (Infections and infestations) | 1
Hepatitis E (Infections and infestations) | 1
Herpes zoster ophthalmic (Infections and infestations) | 1
Incision site cellulitis (Infections and infestations) | 1
Incision site infection (Infections and infestations) | 1
Infected bites (Infections and infestations) | 1
Infected skin ulcer (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Keratitis herpetic (Infections and infestations) | 1
Klebsiella sepsis (Infections and infestations) | 1
Lobar pneumonia (Infections and infestations) | 1
Meningitis aseptic (Infections and infestations) | 1
Mycobacterium avium complex infection (Infections and infestations) | 1
Nasal abscess (Infections and infestations) | 1
Neutropenic sepsis (Infections and infestations) | 1
Osteomyelitis chronic (Infections and infestations) | 1
Paronychia (Infections and infestations) | 1
Parotitis (Infections and infestations) | 1
Perineal infection (Infections and infestations) | 1
Periorbital cellulitis (Infections and infestations) | 1
Peritoneal abscess (Infections and infestations) | 1
Peritonsillar abscess (Infections and infestations) | 1
Pharyngitis streptococcal (Infections and infestations) | 1
Pneumococcal sepsis (Infections and infestations) | 1
Pneumonia bacterial (Infections and infestations) | 1
Pneumonia blastomyces (Infections and infestations) | 1
Pneumonia viral (Infections and infestations) | 1
Post procedural cellulitis (Infections and infestations) | 1
Prostatic abscess (Infections and infestations) | 1
Proteus infection (Infections and infestations) | 1
Pseudomonal bacteraemia (Infections and infestations) | 1
Pseudomonas infection (Infections and infestations) | 1
Psoas abscess (Infections and infestations) | 1
Pyelonephritis acute (Infections and infestations) | 1
Rectal abscess (Infections and infestations) | 1
Renal abscess (Infections and infestations) | 1
Sialoadenitis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Staphylococcal sepsis (Infections and infestations) | 1
Streptococcal sepsis (Infections and infestations) | 1
Systemic candida (Infections and infestations) | 1
Tongue abscess (Infections and infestations) | 1
Tracheitis (Infections and infestations) | 1
Tuberculosis (Infections and infestations) | 1
Varicella (Infections and infestations) | 1
Viral diarrhoea (Infections and infestations) | 1
Wound infection bacterial (Infections and infestations) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 8
Humerus fracture (Injury, poisoning and procedural complications) | 7
Femur fracture (Injury, poisoning and procedural complications) | 5
Pelvic fracture (Injury, poisoning and procedural complications) | 5
Femoral neck fracture (Injury, poisoning and procedural complications) | 4
Joint dislocation (Injury, poisoning and procedural complications) | 4
Upper limb fracture (Injury, poisoning and procedural complications) | 4
Wound dehiscence (Injury, poisoning and procedural complications) | 4
Laceration (Injury, poisoning and procedural complications) | 3
Lower limb fracture (Injury, poisoning and procedural complications) | 3
Spinal compression fracture (Injury, poisoning and procedural complications) | 3
Comminuted fracture (Injury, poisoning and procedural complications) | 2
Foot fracture (Injury, poisoning and procedural complications) | 2
Incisional hernia (Injury, poisoning and procedural complications) | 2
Intentional overdose (Injury, poisoning and procedural complications) | 2
Meniscus injury (Injury, poisoning and procedural complications) | 2
Overdose (Injury, poisoning and procedural complications) | 2
Postoperative ileus (Injury, poisoning and procedural complications) | 2
Postoperative wound complication (Injury, poisoning and procedural complications) | 2
Procedural pain (Injury, poisoning and procedural complications) | 2
Radius fracture (Injury, poisoning and procedural complications) | 2
Seroma (Injury, poisoning and procedural complications) | 2
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 2
Tibia fracture (Injury, poisoning and procedural complications) | 2
Ulna fracture (Injury, poisoning and procedural complications) | 2
Accidental overdose (Injury, poisoning and procedural complications) | 1
Bone fragmentation (Injury, poisoning and procedural complications) | 1
Burns second degree (Injury, poisoning and procedural complications) | 1
Carotid artery restenosis (Injury, poisoning and procedural complications) | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 10
Contusion (Injury, poisoning and procedural complications) | 1
Face injury (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Fracture displacement (Injury, poisoning and procedural complications) | 1
Head injury (Injury, poisoning and procedural complications) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Joint injury (Injury, poisoning and procedural complications) | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1
Multiple fractures (Injury, poisoning and procedural complications) | 1
Multiple injuries (Injury, poisoning and procedural complications) | 1
Patella fracture (Injury, poisoning and procedural complications) | 1
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 1
Post-traumatic pain (Injury, poisoning and procedural complications) | 1
Pubis fracture (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Skull fracture (Injury, poisoning and procedural complications) | 1
Spinal column injury (Injury, poisoning and procedural complications) | 1
Spinal cord injury (Injury, poisoning and procedural complications) | 1
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Synovial rupture (Injury, poisoning and procedural complications) | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 1
Tracheostomy malfunction (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Carcinoid tumour of the gastrointestinal tract (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Diffuse large b-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Lung adenocarcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Lung adenocarcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Lung squamous cell carcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Astrocytoma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Basosquamous carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Benign renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder transitional cell carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dermatofibrosarcoma protuberans (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Fibrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastrointestinal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Intraductal papillary mucinous neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung adenocarcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung squamous cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung squamous cell carcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant anorectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Nasal cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ocular cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian epithelial cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Post transplant lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Sarcoma uterus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Spindle cell sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma of pharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Diverticular perforation (Gastrointestinal disorders) | 11
Abdominal pain (Gastrointestinal disorders) | 6
Gastritis (Gastrointestinal disorders) | 5
Pancreatitis (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 4
Colitis (Gastrointestinal disorders) | 3
Crohn's disease (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 3
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3
Irritable bowel syndrome (Gastrointestinal disorders) | 3
Large intestine perforation (Gastrointestinal disorders) | 3
Small intestinal obstruction (Gastrointestinal disorders) | 3
Abdominal pain upper (Gastrointestinal disorders) | 2
Colitis ischaemic (Gastrointestinal disorders) | 2
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 2
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 2
Gastric ulcer (Gastrointestinal disorders) | 2
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 2
Gastritis erosive (Gastrointestinal disorders) | 2
Haemorrhoids (Gastrointestinal disorders) | 2
Ileus (Gastrointestinal disorders) | 2
Mallory-weiss syndrome (Gastrointestinal disorders) | 2
Abdominal adhesions (Gastrointestinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal wall haematoma (Gastrointestinal disorders) | 1
Anal fissure (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Colitis ulcerative (Gastrointestinal disorders) | 1
Diverticulum (Gastrointestinal disorders) | 1
Diverticulum intestinal (Gastrointestinal disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Enterocutaneous fistula (Gastrointestinal disorders) | 1
Erosive duodenitis (Gastrointestinal disorders) | 1
Food poisoning (Gastrointestinal disorders) | 1
Gastric disorder (Gastrointestinal disorders) | 1
Gastric perforation (Gastrointestinal disorders) | 1
Gastrointestinal erosion (Gastrointestinal disorders) | 1
Gastrointestinal necrosis (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Ileal perforation (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 1
Intussusception (Gastrointestinal disorders) | 1
Large intestinal ulcer (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Oedematous pancreatitis (Gastrointestinal disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Peptic ulcer perforation (Gastrointestinal disorders) | 1
Poor dental condition (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Small intestinal perforation (Gastrointestinal disorders) | 1
Stomatitis haemorrhagic (Gastrointestinal disorders) | 1
Umbilical hernia (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 25
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 7
Foot deformity (Musculoskeletal and connective tissue disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 4
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 4
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 4
Bursitis (Musculoskeletal and connective tissue disorders) | 3
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 3
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 3
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 2
Synovitis (Musculoskeletal and connective tissue disorders) | 2
Acquired claw toe (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Arthrofibrosis (Musculoskeletal and connective tissue disorders) | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1
Fistula (Musculoskeletal and connective tissue disorders) | 1
Fracture malunion (Musculoskeletal and connective tissue disorders) | 1
Joint contracture (Musculoskeletal and connective tissue disorders) | 1
Joint instability (Musculoskeletal and connective tissue disorders) | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 1
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 1
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1
Scoliosis (Musculoskeletal and connective tissue disorders) | 1
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1
Myocardial infarction (Cardiac disorders) | 16
Atrial fibrillation (Cardiac disorders) | 13
Angina pectoris (Cardiac disorders) | 9
Acute myocardial infarction (Cardiac disorders) | 8
Cardiac failure congestive (Cardiac disorders) | 6
Myocardial ischaemia (Cardiac disorders) | 6
Cardiac failure (Cardiac disorders) | 5
Coronary artery disease (Cardiac disorders) | 4
Arrhythmia (Cardiac disorders) | 2
Atrioventricular block complete (Cardiac disorders) | 2
Coronary artery occlusion (Cardiac disorders) | 2
Coronary artery stenosis (Cardiac disorders) | 2
Tachycardia (Cardiac disorders) | 2
Angina unstable (Cardiac disorders) | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 1
Atrial tachycardia (Cardiac disorders) | 1
Atrioventricular block second degree (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure chronic (Cardiac disorders) | 1
Congestive cardiomyopathy (Cardiac disorders) | 1
Diastolic dysfunction (Cardiac disorders) | 1
Mitral valve incompetence (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Stress cardiomyopathy (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Ventricular extrasystoles (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 9
Syncope (Nervous system disorders) | 6
Cerebrovascular accident (Nervous system disorders) | 5
Carotid artery stenosis (Nervous system disorders) | 4
Sciatica (Nervous system disorders) | 3
Cerebral infarction (Nervous system disorders) | 2
Cerebral ischaemia (Nervous system disorders) | 2
Headache (Nervous system disorders) | 2
Intracranial aneurysm (Nervous system disorders) | 2
Ischaemic stroke (Nervous system disorders) | 2
Transient global amnesia (Nervous system disorders) | 2
Viith nerve paralysis (Nervous system disorders) | 2
Aphasia (Nervous system disorders) | 1
Balance disorder (Nervous system disorders) | 1
Carotid artery occlusion (Nervous system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 1
Dementia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Facial neuralgia (Nervous system disorders) | 1
Grand mal convulsion (Nervous system disorders) | 1
Haemorrhagic stroke (Nervous system disorders) | 1
Hypoglycaemic coma (Nervous system disorders) | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1
Intercostal neuralgia (Nervous system disorders) | 1
Ischaemic cerebral infarction (Nervous system disorders) | 1
Lacunar infarction (Nervous system disorders) | 1
Lumbar radiculopathy (Nervous system disorders) | 1
Meralgia paraesthetica (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Migraine with aura (Nervous system disorders) | 1
Monoparesis (Nervous system disorders) | 1
Multiple sclerosis relapse (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Normal pressure hydrocephalus (Nervous system disorders) | 1
Parkinson's disease (Nervous system disorders) | 1
Perineurial cyst (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Ruptured cerebral aneurysm (Nervous system disorders) | 1
Spinal claudication (Nervous system disorders) | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1
Thalamus haemorrhage (Nervous system disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 15
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 7
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 5
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 3
Asthma (Respiratory, thoracic and mediastinal disorders) | 3
Rheumatoid lung (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2
Acute interstitial pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 1
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Deep vein thrombosis (Vascular disorders) | 14
Hypertension (Vascular disorders) | 8
Aortic aneurysm (Vascular disorders) | 4
Haematoma (Vascular disorders) | 2
Hypertensive crisis (Vascular disorders) | 2
Orthostatic hypotension (Vascular disorders) | 2
Phlebitis (Vascular disorders) | 2
Aortic stenosis (Vascular disorders) | 1
Arteriosclerosis (Vascular disorders) | 1
Arteritis (Vascular disorders) | 1
Essential hypertension (Vascular disorders) | 1
Hypovolaemic shock (Vascular disorders) | 1
Peripheral vascular disorder (Vascular disorders) | 1
Post thrombotic syndrome (Vascular disorders) | 1
Thrombosed varicose vein (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 1
Vascular rupture (Vascular disorders) | 1
Non-cardiac chest pain (General disorders) | 11
Device dislocation (General disorders) | 6
Chest pain (General disorders) | 3
Multi-organ failure (General disorders) | 3
Surgical failure (General disorders) | 3
Death (General disorders) | 2
Impaired healing (General disorders) | 2
Cyst (General disorders) | 1
Drug withdrawal syndrome (General disorders) | 1
Effusion (General disorders) | 1
Oedema peripheral (General disorders) | 1
Sudden death (General disorders) | 1
Systemic inflammatory response syndrome (General disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 12
Renal failure acute (Renal and urinary disorders) | 7
Calculus ureteric (Renal and urinary disorders) | 4
Renal failure (Renal and urinary disorders) | 3
Calculus urinary (Renal and urinary disorders) | 2
Hydronephrosis (Renal and urinary disorders) | 1
Incontinence (Renal and urinary disorders) | 1
Mesangioproliferative glomerulonephritis (Renal and urinary disorders) | 1
Obstructive uropathy (Renal and urinary disorders) | 1
Postrenal failure (Renal and urinary disorders) | 1
Renal mass (Renal and urinary disorders) | 1
Ovarian cyst (Reproductive system and breast disorders) | 4
Uterine prolapse (Reproductive system and breast disorders) | 4
Menorrhagia (Reproductive system and breast disorders) | 2
Adnexa uteri cyst (Reproductive system and breast disorders) | 1
Adnexa uteri mass (Reproductive system and breast disorders) | 1
Cervical dysplasia (Reproductive system and breast disorders) | 1
Cervical polyp (Reproductive system and breast disorders) | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 1
Endometriosis (Reproductive system and breast disorders) | 1
Fibrocystic breast disease (Reproductive system and breast disorders) | 1
Postmenopausal haemorrhage 1 (Reproductive system and breast disorders) | 1
Prostatitis (Reproductive system and breast disorders) | 1
Uterine fibrosis (Reproductive system and breast disorders) | 1
Uterine polyp (Reproductive system and breast disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 10
Cholecystitis (Hepatobiliary disorders) | 4
Biliary colic (Hepatobiliary disorders) | 2
Cholecystitis acute (Hepatobiliary disorders) | 2
Bile duct stone (Hepatobiliary disorders) | 1
Cholestasis (Hepatobiliary disorders) | 1
Hepatic steatosis (Hepatobiliary disorders) | 1
Ischaemic hepatitis (Hepatobiliary disorders) | 1
Depression (Psychiatric disorders) | 4
Completed suicide (Psychiatric disorders) | 2
Mental status changes (Psychiatric disorders) | 2
Suicide attempt (Psychiatric disorders) | 2
Abnormal behaviour (Psychiatric disorders) | 1
Alcohol abuse (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 1
Bipolar disorder (Psychiatric disorders) | 1
Bipolar I disorder (Psychiatric disorders) | 1
Conversion disorder (Psychiatric disorders) | 1
Drug dependence (Psychiatric disorders) | 1
Schizophrenia, paranoid type (Psychiatric disorders) | 1
Somatoform disorder neurologic (Psychiatric disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 8
Leukopenia (Blood and lymphatic system disorders) | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 2
Pancytopenia (Blood and lymphatic system disorders) | 2
Anaemia megaloblastic (Blood and lymphatic system disorders) | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 2
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 2
Dry gangrene (Skin and subcutaneous tissue disorders) | 1
Mucocutaneous rash (Skin and subcutaneous tissue disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 3
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1
Cataract (Eye disorders) | 3
Angle closure glaucoma (Eye disorders) | 1
Corneal perforation (Eye disorders) | 1
Retinal artery occlusion (Eye disorders) | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 4
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
Anaphylactic reaction (Immune system disorders) | 2
Allergy to arthropod sting (Immune system disorders) | 1
Anaphylactic shock (Immune system disorders) | 1
Hypoacusis (Ear and labyrinth disorders) | 1
Sudden hearing loss (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Goitre (Endocrine disorders) | 2
Thyroid cyst (Endocrine disorders) | 1
Arnold-chiari malformation (Congenital, familial and genetic disorders) | 1
Choledochal cyst (Congenital, familial and genetic disorders) | 1
Hepatic enzyme increased (Investigations) | 1
Removal of internal fixation 1 (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=2067)
Upper respiratory tract infection (Infections and infestations) | 616
Nasopharyngitis (Infections and infestations) | 495
Urinary tract infection (Infections and infestations) | 420
Bronchitis (Infections and infestations) | 405
Sinusitis (Infections and infestations) | 326
Influenza (Infections and infestations) | 231
Gastroenteritis (Infections and infestations) | 213
Pharyngitis (Infections and infestations) | 180
Herpes zoster (Infections and infestations) | 129
Cellulitis (Infections and infestations) | 127
Gastroenteritis viral (Infections and infestations) | 122
Diarrhoea (Gastrointestinal disorders) | 358
Nausea (Gastrointestinal disorders) | 261
Dyspepsia (Gastrointestinal disorders) | 189
Abdominal pain upper (Gastrointestinal disorders) | 151
Gastritis (Gastrointestinal disorders) | 149
Abdominal pain (Gastrointestinal disorders) | 120
Vomiting (Gastrointestinal disorders) | 114
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 113
Constipation (Gastrointestinal disorders) | 107
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 322
Back pain (Musculoskeletal and connective tissue disorders) | 294
Arthralgia (Musculoskeletal and connective tissue disorders) | 201
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 131
Pain in extremity (Musculoskeletal and connective tissue disorders) | 131
Bursitis (Musculoskeletal and connective tissue disorders) | 117
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 113
Hypertension (Vascular disorders) | 411
Headache (Nervous system disorders) | 289
Dizziness (Nervous system disorders) | 161
Cough (Respiratory, thoracic and mediastinal disorders) | 199
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 115
Oedema peripheral (General disorders) | 183
Fatigue (General disorders) | 128
Insomnia (Psychiatric disorders) | 136
Depression (Psychiatric disorders) | 122
Transaminases increased (Investigations) | 136
Alanine aminotransferase increased (Investigations) | 111
Rash (Skin and subcutaneous tissue disorders) | 181
Hypercholesterolaemia (Metabolism and nutrition disorders) | 170
Contusion (Injury, poisoning and procedural complications) | 149

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.